CLINICAL TRIAL: NCT06634082
Title: Total Extraperitoneal Approach in Orthopedic Surgery (O-TEP); Preliminary Clinical Outcomes of Symphysial Plating in Fifteen Cases: A Case Series'
Brief Title: Total Extraperitoneal Approach in Orthopedic Surgery
Status: Completed | Type: Observational
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Vedat Öztürk, Specialist Doctor in Orthopedics and Traumatology, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Other Study IDs: 2023/299
Record Dates: First submitted 2024-10-06; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Pubic Symphysis Diastasis
Keywords: pubic symphysis diastasis; pelvic ring injury; orthopedic total extraperitoneal approach (O-TEP); endoscopy
MeSH Terms: conditions — Pubic Symphysis Diastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- O-TEP Symphysial Plating Cohort: This cohort consists of 15 patients with pubic symphysis diastasis (PSD) who underwent total extraperitoneal endoscopic symphysial plating (O-TEP) between March 2022 and May 2024. The interventions include a minimally invasive plating procedure aimed at evaluating clinical outcomes, such as postoperative pain, functional recovery, and complications

SUMMARY:
The goal of this retrospective observational study is to evaluate the preliminary clinical and functional outcomes of total extraperitoneal approach (O-TEP) symphysial plating in patients with pubic symphysis diastasis (PSD). The study involved 15 patients (90% male, mean age 40) treated between March 2022 and May 2024.

The main questions it aims to answer are:

What are the clinical outcomes (e.g., VAS scores, Iowa Pelvic Scores, Majeed scores) following O-TEP symphysial plating? What are the surgical outcomes, including operating time, blood loss, and complications, associated with this minimally invasive technique?

Participants underwent:

Total extraperitoneal endoscopic symphysial plating, with follow-up assessments including postoperative pain scores, radiographs, and functional outcome evaluations using the Iowa Pelvic and Majeed scores.

Researchers will analyze the outcomes to see if this approach offers advantages over traditional open surgery, potentially reducing complications and improving recovery in PSD patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with pubic symphysis diastasis (PSD).
* Patients who underwent total extraperitoneal endoscopic symphysial plating (O-TEP) between March 2022 and May 2024.
* Patients with a follow-up period of at least 12 months.
* Patients who provided informed consent for the surgical procedure and the study.

Exclusion Criteria:

* Patients who required conversion to open surgery during the procedure (e.g., due to pneumoperitoneum).
* Patients with a follow-up period of less than 12 months.
* Patients with incomplete clinical or radiological data.
* Patients with contraindications to endoscopic surgery.
* Patients who did not provide informed consent for the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study population consists of patients aged 18-65 years who were diagnosed with pubic symphysis diastasis (PSD) and underwent total extraperitoneal endoscopic symphysial plating (O-TEP) at a Level 1 trauma center between March 2022 and May 2024. Patients included had a minimum follow-up period of 12 months and provided informed consent for the procedure and study participation.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Operating Time | 24 hours (after surgical procedure)
  Time taken to complete the surgical procedure.
Intraoperative Blood Loss | 24 hours (after surgical procedure)
  Amount of blood lost during the surgical procedure.

SECONDARY OUTCOMES:
Postoperative Pain (VAS Scores) | until the final follow-up (12 to 25 months)
  The VAS is scored from 0 to 10, where 0 represents no pain and 10 represents the worst imaginable pain.
Hospital Stay Duration | From the day of surgery until discharge (typically 2 to 4 days). Unit of Measure: Days
  The total number of days the patient stays in the hospital from the day of surgery until discharge.
Complications | From the day of surgery until the final follow-up (12 to 25 months). Unit of Measure: Number of patients with complications.
  Any postoperative complications, including infection, implant failure, or the need for revision surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Bakırköy Dr. Sadi Konuk Training and Research Hospital, Department of Orthopedics and Traumatology, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wake BL, McCormack K, Fraser C, Vale L, Perez J, Grant AM. Transabdominal pre-peritoneal (TAPP) vs totally extraperitoneal (TEP) laparoscopic techniques for inguinal hernia repair. Cochrane Database Syst Rev. 2005 Jan 25;2005(1):CD004703. doi: 10.1002/14651858.CD004703.pub2. PMID 15674961
- [Background] Ozturk V, Bilgili MG. Combining Innovative Techniques: Total Extraperitoneal Approach in Orthopedic Surgery (O-TEP) and Percutaneous Both Column Screw (BCS) Fixation Technique in a Geriatric Acetabular Fracture Case. Z Orthop Unfall. 2025 Aug;163(4):361-367. doi: 10.1055/a-2370-0086. Epub 2024 Aug 13. PMID 39137893
- [Background] Vinet M, Moullac D, David G, Segalen T, Lucas C, Dubrana F, Letissier H, Di Francia R. Laparoscopic treatment of fourteen cases of pelvic ring disruption: a case series. Int Orthop. 2024 Jul;48(7):1859-1869. doi: 10.1007/s00264-024-06170-z. Epub 2024 Apr 18. PMID 38634937
- See also: Related Info — https://link.springer.com/article/10.1007/s00264-024-06213-5